CLINICAL TRIAL: NCT00265733
Title: Phase II Trial of CT-2103 (Xyotax™) With Capecitabine as First-Line Chemotherapy for Patients With Metastatic Breast Cancer
Brief Title: Paclitaxel Poliglumex and Capecitabine in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0437; NCI-2012-02683 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000456449 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: male breast cancer; recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Capecitabine; paclitaxel poliglumex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- paclitaxel + capecitabine (Experimental): Patients receive paclitaxel poliglumex IV (CT-2103; Xyotax™) over 10-20 minutes on day 1 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  After completion of study treatment, patients are followed every 6 months for up to 5 years.
  Interventions: Drug: capecitabine; Drug: paclitaxel poliglumex

INTERVENTIONS:
Drug: capecitabine
Drug: paclitaxel poliglumex

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel poliglumex and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving paclitaxel poliglumex together with capecitabine works in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the tumor response rate and adverse event profile in patients with metastatic, HER2 negative breast cancer treated with paclitaxel poliglumex (CT-2103; Xyotax™) and capecitabine.
* Examine the distributions of disease-free progression times and survival times in these patients.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel poliglumex IV (CT-2103; Xyotax™) over 10-20 minutes on day 1 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologic or cytologic confirmation of breast cancer with clinical evidence of metastatic disease

  * No bone metastases as the only evidence of metastasis
* Measurable disease, defined as at least one measurable lesion

  * No non-measurable disease, defined as all other lesions, including small lesions (longest diameter < 2.0 cm) and truly non-measurable lesions, which include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* No known brain metastasis
* HER2 negative disease by immunohistochemistry and/or fluorescent in situ hybridization
* Diagnostic tissue and operative and pathology reports from breast cancer diagnosis and/or diagnosis of metastatic breast cancer must be available
* Hormone receptor status

  * Not specified

PATIENT CHARACTERISTICS:

* Males or females are eligible
* Menopausal status: not specified
* Life expectancy ≥ 3 months
* ECOG performance status 0 or 1
* Any serum estradiol level allowed
* Hemoglobin > 8.0 g/dL
* Absolute neutrophil count ≥ 1500/mL
* Platelet count ≥ 100,000/mL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* AST and ALT ≤ 2.5 times UNL
* Calcium normal
* Creatinine clearance ≥ 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Women of childbearing potential or their sexual partners must be willing to employ adequate contraception (as determined by the treating physician) for the duration of the study and for 30 days after treatment has ended
* No stage III or IV invasive, non-breast malignancies in ≤ 5 years prior to registration
* No history of allergy or hypersensitivity to capecitabine, paclitaxel, or fluorouracil
* No prior unanticipated severe reaction to fluoropyrimidine therapy
* No known DPD deficiency
* No known, existing uncontrolled coagulopathy
* No uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements
* No lack of physical integrity of the upper gastrointestinal tract, clinically significant malabsorption syndrome, or inability to take oral medication
* No significant medical condition that would make treatment or follow-up on this protocol difficult or problematic, in the opinion of the treating oncologist
* No preexisting neuropathy > grade 0

PRIOR CONCURRENT THERAPY:

* No other concurrent cytotoxic agents, investigational drugs, immunotherapy, radiation therapy or hormonal therapy
* Capecitabine must not be administered together with antiviral drugs
* No concurrent allopurinol, metronidazole, or sorivudine (or its chemically-related analogues, such as brivudine)
* Cimetidine must be discontinued at least 2 weeks prior to start of study treatment and must be avoided while taking capecitabine
* Patients receiving bisphosphonates are eligible for this study
* No prior chemotherapy for metastatic disease
* Prior anthracycline and/or taxane in the neoadjuvant or adjuvant setting allowed if completed ≥ 6 months prior to registration
* Unlimited prior hormonal therapy allowed in the neoadjuvant, adjuvant, or metastatic setting
* No HIV-positive individuals receiving combination anti-retroviral therapy
* No major surgery, chemotherapy, or immunologic therapy ≤ 4 weeks prior to registration
* No radiotherapy ≤ 4 weeks prior to registration, except to a non-target lesion only
* Prior radiation to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed

  * If patient receives single dose radiation for palliation, they may immediately proceed to registration without waiting 4 weeks
* Neoadjuvant and/or adjuvant therapy must be completed > 6 months prior to registration
* No current or recent use (≤ 2 weeks prior to registration) of aspirin, anticoagulants or thrombolytic agents

  * Agents to maintain patency of a vascular access device is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Proportion of confirmed tumor response (complete and partial response) as assessed by RECIST criteria | Up to 5 years

SECONDARY OUTCOMES:
Survival time | Up to 5 years
Time to disease progression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Background] Reinholz MM, Kitzmann KA, Tenner K, Hillman D, Dueck AC, Hobday TJ, Northfelt DW, Moreno-Aspitia A, Roy V, LaPlant B, Allred JB, Stella PJ, Lingle WL, Perez EA. Cytokeratin-19 and mammaglobin gene expression in circulating tumor cells from metastatic breast cancer patients enrolled in North Central Cancer Treatment Group trials, N0234/336/436/437. Clin Cancer Res. 2011 Nov 15;17(22):7183-93. doi: 10.1158/1078-0432.CCR-11-0981. Epub 2011 Oct 5. PMID 21976532
- [Background] Reinholz MM, Kitzmann KA, Hobday TJ, et al.: Cytokeratin-19 (CK19) and mammaglobin (MGB1) gene expression in circulating tumor cells (CTCs) from metastatic breast cancer patients enrolled in the NCCTG trials, N0436 and N0437. [Abstract] J Clin Oncol 27 (Suppl 15): A-11095, 2009.